CLINICAL TRIAL: NCT01458587
Title: A Phase II Study of Photodynamic Therapy (PDT)With LEVULAN® Topical Solution + Blue Light Versus LEVULAN® Topical Solution Vehicle + Blue Light for the Treatment of Actinic Keratoses on the Upper Extremities
Brief Title: Levulan PDT Versus Vehicle for Extremity Actinic Keratoses (AK)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DUSA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP0106
Record Dates: First submitted 2011-10-21; First posted 2011-10-25 (Estimated); Results first posted 2013-02-04 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Keratosis, Actinic
Keywords: Actinic keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALA (Experimental)
  Interventions: Drug: Aminolevulinic Acid PDT (ALA)
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle PDT (VEH)

INTERVENTIONS:
Drug: Aminolevulinic Acid PDT (ALA) — 20% ALA applied to upper extremities for 3 hours prior to 10 J/cm2 blue light
  Other Names: Levulan Kerastick
  Arms: ALA
Drug: Vehicle PDT (VEH) — Levulan Kerastick containing vehicle ingredients only. Vehicle solution applied to upper extremities 3 hours prior to 10 J/cm2 blue light
  Arms: Vehicle

SUMMARY:
The purpose of this study is to determine if Levulan PDT is safe and effective in the treatment of actinic keratoses on the upper arms and hands.

ELIGIBILITY:
Inclusion Criteria:

* At least 4 Grade 1/2 AKs on each upper extremity

Exclusion Criteria:

* Pregnancy
* history of cutaneous photosensitization, porphyria, hypersensitivity to porphyrins or photodermatosis
* lesions suspicious for skin cancer (skin cancer not ruled out by biopsy) or untreated skin cancers within the Treatment Area
* skin pathology or condition which could interfere with the evaluation of the test product or requires the use of interfering topical or systemic therapy
* Subject is immunosuppressed
* unsuccessful outcome from previous ALA-PDT therapy
* currently enrolled in an investigational drug or device study
* has received an investigational drug or been treated with an investigational device within 30 days prior to the initiation of treatment
* known sensitivity to one or more of the vehicle components (ethyl alcohol, isopropyl alcohol, laureth 4, polyethylene glycol)
* use of the following topical preparations on the extremities to be treated:

  * Keratolytics including urea (greater than 5%), alpha hydroxyacids [e.g.glycolic acid, lactic acid, etc. greater than 5%], salicylic acid (greater than 2%) within 2 days of initiation of treatment.
  * Cryotherapy within 2 weeks of initiation of treatment
  * Retinoids, including tazarotene, adapalene, tretinoin, retinol, within 4 weeks of initiation of treatment.
  * Microdermabrasion, laser ablative treatments, ALA-PDT, chemical peels, 5-FU, diclofenac, imiquimod or other topical treatments for AK within 8 weeks of initiation of treatment.
  * Two or more ALA PDT treatments in the past 6 months
* use of systemic retinoid therapy within 6 months of initiation of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Marcus, MD, PhD, Study Director — DUSA Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Therapeutics Clinical Research, San Diego, California
  - Park Avenue Dermatology, PA, Orange Park, Florida
  - DermResearch, Inc, Austin, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was from 28November2011 - 4April2012 at 3 medical clinics in the U.S.
Groups:
- Aminolevulinic Acid: ALA applied to both extremities; one extremity on each subject randomized to occlusion with plastic wrap during the incubation period.
- Vehicle: Vehicle applied to both extremities; one extremity on each subject randomized to occlusion with plastic wrap during the incubation period.
Period: Overall Study
Arm/Group | Aminolevulinic Acid | Vehicle
Started | 35 | 35
Completed | 34 | 35
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aminolevulinic Acid | Vehicle | Total
Number analyzed (Participants) | 35 | 35 | 70
Age Continuous [Mean (Standard Deviation); unit: years] | 62.1 (9.96) | 65.6 (9.30) | 63.8 (9.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 22 | 23 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 35 | 35 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 35 | 35 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Lesion Clearance Rate
Description: Clearance rate for all lesions
Time Frame: Week 12
Population: ITT analysis with LOCF
Measure: Median (Standard Deviation); unit: percentage of lesions cleared
Units Other Than Participants: arms
Groups:
- ALA+OCC: ALA application on one extremity occluded with plastic wrap during the incubation period.
- ALA-OCC: ALA application on one extremity unoccluded during the incubation period.
- VEH+OCC: Vehicle application on one extremity occluded with plastic wrap during the incubation period.
- VEH-OCC: Vehicle application on one extremity unoccluded during the incubation period.
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 35 | 35
Number analyzed (arms) | 35 | 35 | 35 | 35
percentage of lesions cleared | 88.7 (25.1) | 70.0 (31.1) | 16.7 (27.6) | 5.6 (26.8)

2. Secondary Outcome: Lesion Clearance Rate
Time Frame: Week 8
Population: ITT LOCF
Measure: Median (Standard Deviation); unit: percentage of lesions cleared
Units Other Than Participants: arms
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 35 | 35
Number analyzed (arms) | 35 | 35 | 35 | 35
percentage of lesions cleared | 75.0 (34.6) | 47.4 (30.7) | 3.3 (28.7) | 6.3 (25.8)

3. Secondary Outcome: Complete Clearance Rate
Description: proportion of subjects with a count of zero lesions in the treatment area
Time Frame: Week 8
Population: ITT LOCF
Measure: Number; unit: arms 100% cleared
Units Other Than Participants: arms
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 35 | 35
Number analyzed (arms) | 35 | 35 | 35 | 35
arms 100% cleared | 8 | 4 | 0 | 0

4. Secondary Outcome: Complete Clearance Rate
Description: proportion of subjects with a count of zero lesions in the treatment area
Time Frame: Week 12
Population: ITT LOCF
Measure: Number; unit: arms 100% cleared
Units Other Than Participants: arms
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 35 | 35
Number analyzed (arms) | 35 | 35 | 35 | 35
arms 100% cleared | 12 | 7 | 0 | 1

5. Secondary Outcome: Partial Clearance Rate
Description: proportion of subjects with 75% or more reduction in the AK count in the Treatment Area as compared to baseline.
Time Frame: Baseline and Week 8
Population: ITT LOCF
Measure: Number; unit: arms >75% cleared
Units Other Than Participants: arms
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 35 | 35
Number analyzed (arms) | 35 | 35 | 35 | 35
arms >75% cleared | 18 | 5 | 1 | 2

6. Secondary Outcome: Partial Clearance Rate
Description: proportion of subjects with 75% or more reduction in the AK count in the Treatment Area as compared to baseline.
Time Frame: Baseline and Week 12
Population: ITT LOCF
Measure: Number; unit: arms >75% cleared
Units Other Than Participants: arms
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 35 | 35
Number analyzed (arms) | 35 | 35 | 35 | 35
arms >75% cleared | 21 | 15 | 3 | 2

7. Secondary Outcome: Subject Satisfaction Score
Description: Subject satisfaction score
  1. = Excellent (very satisfied)
  2. = Good (moderately satisfied)
  3. = Fair (slightly satisfied)
  4. = Poor (not satisfied at all)
Time Frame: Week 12
Population: ITT
Measure: Number; unit: participants
Units Other Than Participants: arms
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 35 | 35
Number analyzed (arms) | 35 | 35 | 35 | 35
participants
  Very satisfied | 13 | 7 | 3 | 1
  Moderately satisfied | 16 | 14 | 5 | 5
  Slightly satisfied | 3 | 8 | 7 | 9
  Not satisfied | 3 | 6 | 20 | 20

8. Secondary Outcome: Hyperpigmentation at Baseline
Description: HYPERPIGMENTATION SCALE Grade 0 = No hyperpigmentation Grade 1 = Light hyperpigmentation involving small areas Grade 2 = Moderate hyperpigmentation involving small areas; light hyperpigmentation involving moderate areas Grade 3 = Moderate hyperpigmentation involving moderate sized areas; light hyperpigmentation involving large areas; small areas of marked hyperpigmentation Grade 4 = Marked hyperpigmentation involving moderate or large sized areas
Time Frame: Baseline
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  Grade 0 (none) | 5 | 5 | 1 | 1
  Grade 1 (light) | 20 | 19 | 23 | 23
  Grade 2 (moderate - small) | 9 | 10 | 8 | 8
  Grade 3 (moderate - moderate) | 1 | 1 | 3 | 3

9. Secondary Outcome: Hyperpigmentation at Visit 3
Description: as for outcome 8
Time Frame: 2 weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 34 | 35 | 35 | 35
participants
  Grade 0 (none) | 4 | 4 | 1 | 1
  Grade 1 (light) | 19 | 20 | 21 | 21
  Grade 2 (moderate - small) | 9 | 10 | 10 | 10
  Grade 3 (moderate - moderate) | 2 | 1 | 3 | 3

10. Secondary Outcome: Hyperpigmentation at Visit 4
Description: as for outcome 8
Time Frame: 8 weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 34 | 34
participants
  Grade 0 (none) | 2 | 2 | 0 | 0
  Grade 1 (light) | 24 | 21 | 19 | 17
  Grade 2 (moderate - small) | 8 | 11 | 11 | 13
  Grade 3 (moderate - moderate) | 1 | 1 | 4 | 4

11. Secondary Outcome: Hyperpigmentation at Visit 5
Description: as for outcome 8
Time Frame: 12 weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 33 | 33 | 35 | 35
participants
  Grade 0 (none) | 2 | 2 | 0 | 0
  Grade 1 (light) | 25 | 23 | 20 | 20
  Grade 2 (moderate - small) | 6 | 8 | 11 | 11
  Grade 3 (moderate - moderate) | 0 | 0 | 4 | 4

12. Secondary Outcome: Hypopigmentation at Baseline
Description: HYPOPIGMENTATION SCALE Grade 0 = No hypopigmentation Grade 1 = Light hypopigmentation involving small areas Grade 2 = Moderate hypopigmentation involving small areas; light hypopigmentation involving moderate areas Grade 3 = Moderate hypopigmentation involving moderate sized areas; light hypopigmentation involving large areas; small areas of marked hypopigmentation
Time Frame: Baseline
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  Grade 0 (none) | 9 | 9 | 8 | 8
  Grade 1 (light) | 21 | 21 | 24 | 24
  Grade 2 (moderate - small) | 5 | 5 | 2 | 2
  Grade 3 (moderate - moderate) | 0 | 0 | 1 | 1

13. Secondary Outcome: Hypopigmentation at Visit 3
Description: as for outcome 12
Time Frame: 2 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 34 | 35 | 35 | 35
participants
  Grade 0 (none) | 10 | 10 | 7 | 7
  Grade 1 (light) | 20 | 20 | 26 | 26
  Grade 2 (moderate - small) | 4 | 5 | 1 | 1
  Grade 3 (moderate - moderate) | 0 | 0 | 1 | 1

14. Secondary Outcome: Hypopigmentation at Visit 4
Description: as for outcome 12
Time Frame: 8 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 34 | 34
participants
  Grade 0 (none) | 13 | 10 | 9 | 9
  Grade 1 (light) | 18 | 21 | 23 | 23
  Grade 2 (moderate - small) | 3 | 4 | 1 | 1
  Grade 3 (moderate - moderate) | 1 | 0 | 1 | 1

15. Secondary Outcome: Hypopigmentation at Visit 5
Description: as for outcome 12
Time Frame: 12 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 33 | 33 | 35 | 35
participants
  Grade 0 (none) | 10 | 8 | 12 | 11
  Grade 1 (light) | 22 | 24 | 21 | 22
  Grade 2 (moderate - small) | 1 | 1 | 1 | 1
  Grade 3 (moderate - moderate) | 0 | 0 | 1 | 1

16. Secondary Outcome: Erythema at Baseline
Description: Erythema Scale - Grade 0 = None Grade 1 = Minimal - barely perceptible erythema Grade 2 = Mild - predominantly minimal erythema (pink) in the treated area with or without a few isolated areas of more intense erythema Grade 3 = Moderate - predominantly moderate erythema (red) in the treated area with or without a few isolated areas of intense erythema (bright red) Grade 4 = Severe - predominantly intense erythema (bright red) in the treated area with or without a few isolated areas of very intense (fiery red) erythema
Time Frame: Baseline
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  Grade 0 (none) | 10 | 10 | 12 | 12
  Grade 1 (minimal) | 16 | 16 | 13 | 12
  Grade 2 (mild) | 8 | 9 | 9 | 10
  Grade 3 (moderate) | 1 | 0 | 1 | 1
  Grade 4 (severe) | 0 | 0 | 0 | 0

17. Secondary Outcome: Erythema Post-Light Treatment
Description: as for outcome 16
Time Frame: 5 Minutes after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  Grade 0 (none) | 0 | 0 | 4 | 4
  Grade 1 (minimal) | 0 | 4 | 11 | 15
  Grade 2 (mild) | 7 | 19 | 17 | 13
  Grade 3 (moderate) | 21 | 10 | 3 | 3
  Grade 4 (severe) | 7 | 2 | 0 | 0

18. Secondary Outcome: Erythema at Visit 3
Description: as for outcome 16
Time Frame: 2 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  Grade 0 (none) | 0 | 4 | 10 | 10
  Grade 1 (minimal) | 8 | 14 | 15 | 14
  Grade 2 (mild) | 14 | 15 | 9 | 10
  Grade 3 (moderate) | 12 | 2 | 1 | 1
  Grade 4 (severe) | 1 | 0 | 0 | 0

19. Secondary Outcome: Erythema at Visit 4
Description: as for outcome 16
Time Frame: 8 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 34 | 34
participants
  Grade 0 (none) | 7 | 6 | 10 | 11
  Grade 1 (minimal) | 17 | 20 | 16 | 15
  Grade 2 (mild) | 9 | 9 | 7 | 7
  Grade 3 (moderate) | 2 | 0 | 1 | 1
  Grade 4 (severe) | 0 | 0 | 0 | 0

20. Secondary Outcome: Erythema at Visit 5
Description: as for outcome 16
Time Frame: 12 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 33 | 33 | 35 | 35
participants
  Grade 0 (none) | 9 | 7 | 11 | 12
  Grade 1 (minimal) | 7 | 12 | 14 | 14
  Grade 2 (mild) | 16 | 14 | 10 | 9
  Grade 3 (moderate) | 1 | 0 | 0 | 0
  Grade 4 (severe) | 0 | 0 | 0 | 0

21. Secondary Outcome: Edema at Baseline
Description: EDEMA SCALE Grade 0 = None Grade 1 = Minimal - scant, rare edema Grade 2 = Mild - easily seen edema, minimally palpable, involving up to 1/3 of the treatment area Grade 3 = Moderate - easily seen edema and typically palpable, involving between 1/3 to 2/3 of the treatment area Grade 4 = Severe - easily seen edema, indurated in some areas, involving over 2/3 of the treatment area
Time Frame: Baseline
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  Grade 0 (none) | 35 | 35 | 35 | 35
  Grade 1 (minimal) | 0 | 0 | 0 | 0
  Grade 2 (mild) | 0 | 0 | 0 | 0

22. Secondary Outcome: Edema Post-Light Treatment
Description: as for outcome 21
Time Frame: 5 Minutes after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  Grade 0 (none) | 28 | 33 | 34 | 34
  Grade 1 (minimal) | 5 | 2 | 1 | 1
  Grade 2 (mild) | 2 | 0 | 0 | 0

23. Secondary Outcome: Edema at Visit 3
Description: as for outcome 21
Time Frame: 2 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  Grade 0 (none) | 27 | 34 | 35 | 35
  Grade 1 (minimal) | 5 | 1 | 0 | 0
  Grade 2 (mild) | 3 | 0 | 0 | 0

24. Secondary Outcome: Edema at Visit 4
Description: as for outcome 21
Time Frame: 8 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 34 | 34
participants
  Grade 0 (none) | 35 | 35 | 34 | 34
  Grade 1 (minimal) | 0 | 0 | 0 | 0
  Grade 2 (mild) | 0 | 0 | 0 | 0

25. Secondary Outcome: Edema at Visit 5
Description: as for outcome 21
Time Frame: 12 Weeks after PDT #1
Population: ITT
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 33 | 33 | 35 | 35
participants
  Grade 0 (none) | 33 | 33 | 35 | 35
  Grade 1 (minimal) | 0 | 0 | 0 | 0
  Grade 2 (mild) | 0 | 0 | 0 | 0

26. Secondary Outcome: Stinging/Burning at Baseline
Description: STINGING AND BURNING SCALE Grade 0 = None Grade 1 = Minimal, barely perceptible -tolerable and little discomfort Grade 2 = Moderate - tolerable, but causes some discomfort Grade 3 = Severe - very uncomfortable or intolerable
Time Frame: Baseline
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  Grade 0 (none) | 35 | 35 | 35 | 35
  Grade 1 (mild) | 0 | 0 | 0 | 0
  Grade 2 (moderate) | 0 | 0 | 0 | 0
  Grade 3 (severe) | 0 | 0 | 0 | 0

27. Secondary Outcome: Stinging/Burning During Light Treatment
Description: as for outcome 26
Time Frame: During PDT #1
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  Grade 0 (none) | 0 | 0 | 29 | 29
  Grade 1 (mild) | 5 | 20 | 6 | 6
  Grade 2 (moderate) | 21 | 12 | 0 | 0
  Grade 3 (severe) | 9 | 3 | 0 | 0

28. Secondary Outcome: Stinging/Burning Post Light Treatment
Description: as for outcome 26
Time Frame: 5 minutes after PDT #1
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  Grade 0 (none) | 0 | 2 | 30 | 33
  Grade 1 (mild) | 7 | 22 | 5 | 2
  Grade 2 (moderate) | 21 | 10 | 0 | 0
  Grade 3 (severe) | 7 | 1 | 0 | 0

29. Secondary Outcome: Stinging/Burning at Visit 3
Description: as for outcome 26
Time Frame: 2 Weeks after PDT #1
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  Grade 0 (none) | 31 | 35 | 35 | 35
  Grade 1 (mild) | 4 | 0 | 0 | 0
  Grade 2 (moderate) | 0 | 0 | 0 | 0
  Grade 3 (severe) | 0 | 0 | 0 | 0

30. Secondary Outcome: Stinging/Burning at Visit 4
Description: as for outcome 26
Time Frame: 8 Weeks after PDT #1
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 34 | 34
participants
  Grade 0 (none) | 35 | 35 | 34 | 34
  Grade 1 (mild) | 0 | 0 | 0 | 0
  Grade 2 (moderate) | 0 | 0 | 0 | 0
  Grade 3 (severe) | 0 | 0 | 0 | 0

31. Secondary Outcome: Stinging/Burning at Visit 5
Description: as for outcome 26
Time Frame: 12 Weeks after PDT #1
Population: ITT, observed
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 33 | 33 | 35 | 35
participants
  Grade 0 (none) | 33 | 33 | 35 | 35
  Grade 1 (mild) | 0 | 0 | 0 | 0
  Grade 2 (moderate) | 0 | 0 | 0 | 0
  Grade 3 (severe) | 0 | 0 | 0 | 0

32. Secondary Outcome: Scaling and Dryness at Baseline
Description: SCALING AND DRYNESS SCALE Grade 0 = None Grade 1 = Minimal - barely perceptible desquamation Grade 2 = Mild - limited areas of fine desquamation in up to 1/3 of the treatment area Grade 3 = Moderate - fine desquamation involving 1/3 to 2/3 of the treatment area or limited areas of coarser scaling Grade 4 = Severe - coarser scaling involving more than 2/3 of the treatment area or limited areas of very coarse scaling
Time Frame: Baseline
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  Grade 0 (none) | 16 | 16 | 17 | 17
  Grade 1 (minimal) | 15 | 15 | 13 | 13
  Grade 2 (mild) | 2 | 2 | 4 | 4
  Grade 3 (moderate) | 2 | 2 | 1 | 1
  Grade 4 (severe) | 0 | 0 | 0 | 0

33. Secondary Outcome: Scaling and Dryness at Visit 3
Description: as for outcome 32
Time Frame: 2 Weeks Post PDT #1
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  Grade 0 (none) | 3 | 5 | 10 | 11
  Grade 1 (minimal) | 5 | 17 | 20 | 19
  Grade 2 (mild) | 5 | 10 | 3 | 3
  Grade 3 (moderate) | 21 | 3 | 2 | 2
  Grade 4 (severe) | 1 | 0 | 0 | 0

34. Secondary Outcome: Scaling and Dryness at Visit 4
Description: as for outcome 32
Time Frame: 8 Weeks Post PDT #1
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 34 | 34
participants
  Grade 0 (none) | 16 | 17 | 14 | 14
  Grade 1 (minimal) | 14 | 12 | 14 | 14
  Grade 2 (mild) | 4 | 5 | 3 | 3
  Grade 3 (moderate) | 1 | 1 | 3 | 3
  Grade 4 (severe) | 0 | 0 | 0 | 0

35. Secondary Outcome: Scaling and Dryness at Visit 5
Description: as for outcome 32
Time Frame: 12 Weeks Post PDT #1
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 33 | 33 | 35 | 35
participants
  Grade 0 (none) | 18 | 17 | 12 | 12
  Grade 1 (minimal) | 12 | 13 | 17 | 17
  Grade 2 (mild) | 2 | 2 | 5 | 5
  Grade 3 (moderate) | 1 | 1 | 1 | 1
  Grade 4 (severe) | 0 | 0 | 0 | 0

36. Secondary Outcome: OOZING/VESICULATION/CRUSTING at Baseline
Description: OOZING/VESICULATION/CRUSTING Grade 0 = None Grade 1 = Minimal - a single area of oozing, vesiculation or crusting 3 mm diameter or less in size Grade 2 = Mild - two to four areas of oozing, vesiculation or crusting 3 mm diameter or less in size OR a single area larger than 3 mm diameter in size Grade 3 = Moderate - more than a single area of oozing, vesiculation or crusting larger than 3 mm diameter in size or more than four areas of 3 mm diameter or less in size Grade 4 = Severe - any degree of oozing, vesiculation or crusting greater than (3) above
Time Frame: Baseline
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  Grade 0 (none) | 35 | 35 | 35 | 35
  Grade 1 (minimal) | 0 | 0 | 0 | 0
  Grade 2 (mild) | 0 | 0 | 0 | 0
  Grade 3 (moderate) | 0 | 0 | 0 | 0
  Grade 4 (severe) | 0 | 0 | 0 | 0

37. Secondary Outcome: OOZING/VESICULATION/CRUSTING at Visit 3
Description: as for outcome 36
Time Frame: Week 2 after PDT #1
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  Grade 0 (none) | 33 | 34 | 34 | 34
  Grade 1 (minimal) | 1 | 0 | 1 | 1
  Grade 2 (mild) | 0 | 1 | 0 | 0
  Grade 3 (moderate) | 1 | 0 | 0 | 0
  0 | 0 | 0 | 0 | 0

38. Secondary Outcome: OOZING/VESICULATION/CRUSTING at Visit 4
Description: as for outcome 36
Time Frame: 8 Weeks after PDT #1
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 35 | 35 | 34 | 34
participants
  Grade 0 (none) | 35 | 35 | 34 | 34
  Grade 1 (minimal) | 0 | 0 | 0 | 0
  Grade 2 (mild) | 0 | 0 | 0 | 0
  Grade 3 (moderate) | 0 | 0 | 0 | 0
  0 | 0 | 0 | 0 | 0

39. Secondary Outcome: OOZING/VESICULATION/CRUSTING at Visit 5
Description: as for outcome 36
Time Frame: 12 Weeks after PDT #1
Population: ITT observed
Measure: Number; unit: participants
Arm/Group | ALA+OCC | ALA-OCC | VEH+OCC | VEH-OCC
Number analyzed (Participants) | 33 | 33 | 35 | 35
participants
  Grade 0 (none) | 33 | 32 | 35 | 35
  Grade 1 (minimal) | 0 | 1 | 0 | 0
  Grade 2 (mild) | 0 | 0 | 0 | 0
  Grade 3 (moderate) | 0 | 0 | 0 | 0
  0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Aminolevulinic Acid | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 17/35 | 5/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aminolevulinic Acid (N=35) | Vehicle (N=35)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pain (Skin and subcutaneous tissue disorders) | 9 (10) | 0 (0) — PDT Reaction
Itching (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — PDT reaction
Swelling (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — PDT reaction

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication of results from multi-center trial will be made by the Sponsor. If publication is not submitted within 12 months after conclusion of the study, the PI may publish the results from the site individually, subject to compliance with the other terms of the clinical trial agreement, including a requirement that the PI provide a draft of the publication for the sponsor's review 60 days before publication so that sponsor can review the publication for confidential information.